CLINICAL TRIAL: NCT07122037
Title: Mechanical and Sensorial Training in the Olfactive Rehabilitation of Patients With Total Laryngectomy : a Randomized Controlled Study
Brief Title: Mechanical and Sensorial Training in the Olfactive Rehabilitation of Patients With Total Laryngectomy
Acronym: OLFAC-TL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Nève Jean-Gualbert, Medical Doctor, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 52/2021
Record Dates: First submitted 2025-07-24; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Aging; Hyposmia; Total Laryngectomy
Keywords: Anosmia; Hyposmia; Total laryngectomy; Quality of life; Olfactory bulb volume; Sniffin' Sticks Test; NAIM
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAIM + OT (Experimental): Total laryngectomy patients receiving olfactory rehabilitation with NAIM maneuver and olfactory training
  Interventions: Device: DosMedical Smell Training Set; Behavioral: Nasal Airflow Inducing Maneuver
- NAIM (Active Comparator): Total laryngectomy patients receiving olfactory rehabilitation only with the NAIM maneuver
  Interventions: Behavioral: Nasal Airflow Inducing Maneuver

INTERVENTIONS:
Device: DosMedical Smell Training Set — Olfactory training with four different odorants (e.g., rose, eucalyptus, lemon, and cloves) for approximately 10 seconds each, twice a day, in the morning and in the evening
  Arms: NAIM + OT
Behavioral: Nasal Airflow Inducing Maneuver — Repeated generation of an "underpressure" in the oral cavity by simultaneously lowering the jaw, the floor of the mouth the tongue, the base of the tongue and soft palate with securely closed lips. This negative pressure created in the oral cavity generates an airflow through the nose.

SUMMARY:
To assess the efficacy of two olfactory rehabilitation protocols (Nasal Airflow-Inducing Maneuver (NAIM) with or without ol-factory training) on olfactory function (sniffing stick test) and quality of life (questionnaire Self-MOQ and EORTC QLQ-H&N35) in patients with total laryngectomy.

ELIGIBILITY:
Inclusion criteria

* Man or woman over 18 years of age, with no upper age limit
* Patient scheduled to total laryngectomy either for oncological purpose (treatment approved by local tumor board) or for functional purpose (se-vere chronic inhalation)
* Capacity to understand and voluntarily sign an informed consent form. Exclusion criteria
* Insufficient French language skills.
* Preexistent anosmia (Sniffin' Stick test score <16/48)
* Contraindications to MRI imaging (e.g., metallic foreign bodies, claustro-phobia…)
* Severe chronic rhinosinusitis with polyps (Davos score 3 or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Olfactory function | From total laryngectomy to the end of olfactory rehabilitation at 1 year
  Prospectively assess the effect on olfactory function of adding olfactory training to a Nasal Airflow-Inducing Maneuver (NAIM) rehabilitation protocol after total laryngectomy.
  Olfactory function was measured with the Sniffin' Sticks Test battery before surgery and at 1, 3, 6, and 12 months after surgery. According to normative data, hyposmia was defined as TDI scores ranging from 16.25 to 30.5, while functional anosmia was classified as a TDI score of 16 or below.
Olfactory-related quality of life | From total laryngectomy to the end of olfactory rehabilitation at 1 year
  Prospectively assess the effect on olfactory-related quality of life of adding olfactory training to a Nasal Airflow-Inducing Maneuver (NAIM) rehabilitation protocol after total laryngectomy.
  Participants assessed their smell-related quality of life using the validated Self-reported Mini Olfactory Questionnaire (Self-MOQ) before surgery and at 1, 3, 6, and 12 months after surgery. Additionally, the EORTC QLQ-H&N35 questionnaire was used, specifically its senses scale, with scoring conducted according to the EORTC scoring manual. A higher score indicated greater olfactory dysfunction in both questionnaires.

SECONDARY OUTCOMES:
Olfactory bulb volume | Pre-operatively and 6 months after total laryngectomy
  Investigate the impact of olfactory rehabilitation on the olfactory bulb volume after laryngectomy.
  Olfactory bulb volume was measured on brain magnetic resonance imaging focusing on the olfactory bulb conducted preoperatively and six months after total laryngectory using a 3 Tesla system. Olfactory bulb volumes were measured bilaterally using coronal T2-weighted images with 2 mm-thick slices and no gaps.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU UCL Namur Site Godinne, Yvoir, Belgium